CLINICAL TRIAL: NCT01854047
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Study to Evaluate Dupilumab in Patients With Moderate to Severe Uncontrolled Asthma
Brief Title: An Evaluation of Dupilumab in Patients With Moderate to Severe Uncontrolled Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DRI12544; 2013-000856-16 (EudraCT Number); U1111-1138-3962 (Other: UTN)
Record Dates: First submitted 2013-05-10; First posted 2013-05-15 (Estimated); Results first posted 2017-06-02 (Actual); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — dupilumab; Albuterol; Levalbuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Dupilumab 300 mg q2w (Experimental): 2 subcutaneous injections of Dupilumab 300 mg (for a total of 600 mg) as a loading dose on Day 1 (Week 1), followed by a single 300 mg injection q2w from Week 2 to Week 22 added to stable inhaled corticosteroid/ long-acting beta-agonist (ICS/LABA) therapy. Salbutamol/albuterol or Levosalbutamol/levalbuterol was given as reliever medication.
  Interventions: Drug: Dupilumab; Drug: ICS/LABA therapy; Drug: Salbutamol/albuterol; Drug: Levosalbutamol/levalbuterol
- Dupilumab 200 mg q2w (Experimental): 2 subcutaneous injections of Dupilumab 200 mg (for a total of 400 mg) as a loading dose on Day 1 (Week 1), followed by a single 200 mg injection q2w from Week 2 to Week 22 added to stable ICS/LABA therapy. Salbutamol/albuterol or Levosalbutamol/levalbuterol was given as reliever medication.
  Interventions: Drug: Dupilumab; Drug: ICS/LABA therapy; Drug: Salbutamol/albuterol; Drug: Levosalbutamol/levalbuterol
- Dupilumab 300 mg q4w (Experimental): 2 subcutaneous injections of Dupilumab 300 mg (for a total of 600 mg) as a loading dose on Day 1 (Week 1) followed by a Placebo alternating with single 300 mg injection of Dupilumab q2w from Week 2 to Week 22 added to stable ICS/LABA therapy. Salbutamol/albuterol or Levosalbutamol/levalbuterol was given as reliever medication.
  Interventions: Drug: Dupilumab; Drug: placebo; Drug: ICS/LABA therapy; Drug: Salbutamol/albuterol; Drug: Levosalbutamol/levalbuterol
- Dupilumab 200 mg q4w (Experimental): 2 subcutaneous injections of Dupilumab 200 mg (for a total of 400 mg) as a loading dose on Day 1 (Week 1) followed by a Placebo alternating with single 200 mg injection of Dupilumab q2w from Week 2 to Week 22 added to stable ICS/LABA therapy. Salbutamol/albuterol or Levosalbutamol/levalbuterol was given as reliever medication.
  Interventions: Drug: Dupilumab; Drug: placebo; Drug: ICS/LABA therapy; Drug: Salbutamol/albuterol; Drug: Levosalbutamol/levalbuterol
- Placebo q2w (Placebo Comparator): 2 subcutaneous injections of Placebo (for Dupilumab) as a loading dose on Day 1 (Week 1) followed by a single injection q2w from Week 2 to Week 22 added to stable ICS/LABA therapy. Salbutamol/albuterol or Levosalbutamol/levalbuterol was given as reliever medication.
  Interventions: Drug: placebo; Drug: ICS/LABA therapy; Drug: Salbutamol/albuterol; Drug: Levosalbutamol/levalbuterol

INTERVENTIONS:
Drug: Dupilumab — Solution for injection, Subcutaneous injection
  Other Names: SAR231893; REGN668
  Arms: Dupilumab 200 mg q2w; Dupilumab 200 mg q4w; Dupilumab 300 mg q2w; Dupilumab 300 mg q4w
Drug: placebo — Solution for injection, Subcutaneous injection
  Arms: Dupilumab 200 mg q4w; Dupilumab 300 mg q4w; Placebo q2w
Drug: ICS/LABA therapy — Oral inhalation, Prior therapy with Mometasone furoate /formoterol, budesonide / formoterol, or fluticasone propionate / salmeterol continued at stable dose
Drug: Salbutamol/albuterol — Oral inhalation as needed
Drug: Levosalbutamol/levalbuterol — Oral inhalation as needed

SUMMARY:
Primary Objective:

To evaluate the efficacy of different doses and regimens of dupilumab in participants with moderate to severe uncontrolled asthma.

Secondary Objective:

To evaluate different doses and regimens of dupilumab in participants with moderate to severe uncontrolled asthma, with regard to:

* Safety and tolerability
* Dupilumab systemic exposure and anti-drug antibodies

DETAILED DESCRIPTION:
Total duration per participant of approximately 43 weeks including a screening period (14-21 days), a randomized treatment period (24 weeks), and a post-treatment period (16 weeks).

ELIGIBILITY:
Inclusion criteria:

Participants with a physician diagnosis of moderate to severe, uncontrolled asthma for >=12 months, based on the Global Initiative for Asthma (GINA) 2009 Guidelines and:

* Existing treatment with moderate or high-dose inhaled corticosteroid / long-acting beta-2 agonist
* Forced expiratory volume (FEV1) 40 to 80% of predicted normal
* Asthma Control Questionnaire, 5-question version (ACQ-5) score >=1.5
* Reversibility of at least 12% and 200 mL in forced expiratory volume (FEV1)
* Had experienced, within prior year: hospitalization, emergency or urgent care visit or systemic corticosteroid treatment for worsening asthma

Exclusion criteria:

* Participants <18 years
* Chronic obstructive pulmonary disease (COPD) or other lung diseases (eg, emphysema, idiopathic pulmonary fibrosis, Churg-Strauss syndrome, allergic bronchopulmonary aspergillosis) which impaired pulmonary function tests
* Chest X-ray within 12 months of screening visit or at screening visit with clinically significant findings of lung disease(s) other than asthma
* Current smoker or cessation of smoking within 6 months prior to Visit 1
* Previous smoker with a smoking history >10 pack-years

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 776 (Actual)
Dates: Start 2013-06; Primary Completion 2014-11 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (201):
- United States (50):
  - Investigational Site Number 840050, Fullerton, California
  - Investigational Site Number 840041, Huntington Beach, California
  - Investigational Site Number 840019, Los Angeles, California
  - Investigational Site Number 840029, Los Angeles, California
  - Investigational Site Number 840022, Los Angeles, California
  - Investigational Site Number 840013, Mission Viejo, California
  - Investigational Site Number 840044, Newport Beach, California
  - Investigational Site Number 840007, Riverside, California
  - Investigational Site Number 840014, Rolling Hills Estates, California
  - Investigational Site Number 840036, San Jose, California
  - Investigational Site Number 840032, Colorado Springs, Colorado
  - Investigational Site Number 840040, Colorado Springs, Colorado
  - Investigational Site Number 840043, Denver, Colorado
  - Investigational Site Number 840006, Denver, Colorado
  - Investigational Site Number 840024, Denver, Colorado
  - Investigational Site Number 840027, Daytona Beach, Florida
  - Investigational Site Number 840039, Miami, Florida
  - Investigational Site Number 840048, Albany, Georgia
  - Investigational Site Number 840026, River Forest, Illinois
  - Investigational Site Number 840053, Evansville, Indiana
  - Investigational Site Number 840017, Louisville, Kentucky
  - Investigational Site Number 840030, Owensboro, Kentucky
  - Investigational Site Number 840028, Baltimore, Maryland
  - Investigational Site Number 840052, Wheaton, Maryland
  - Investigational Site Number 840045, North Dartmouth, Massachusetts
  - Investigational Site Number 840046, Novi, Michigan
  - Investigational Site Number 840051, Novi, Michigan
  - Investigational Site Number 840018, Minneapolis, Minnesota
  - Investigational Site Number 840002, St Louis, Missouri
  - Investigational Site Number 840003, St Louis, Missouri
  - Investigational Site Number 840037, Missoula, Montana
  - Investigational Site Number 840004, Papillion, Nebraska
  - Investigational Site Number 840011, Princeton, New Jersey
  - Investigational Site Number 840016, Rochester, New York
  - Investigational Site Number 840025, Cincinnati, Ohio
  - Investigational Site Number 840015, Cincinnati, Ohio
  - Investigational Site Number 840020, Cincinnati, Ohio
  - Investigational Site Number 840001, Oklahoma City, Oklahoma
  - Investigational Site Number 840031, Lake Oswego, Oregon
  - Investigational Site Number 840034, Medford, Oregon
  - Investigational Site Number 840042, Philadelphia, Pennsylvania
  - Investigational Site Number 840010, Pittsburgh, Pennsylvania
  - Investigational Site Number 840009, Upland, Pennsylvania
  - Investigational Site Number 840021, Spartanburg, South Carolina
  - Investigational Site Number 840023, Dallas, Texas
  - Investigational Site Number 840005, El Paso, Texas
  - Investigational Site Number 840008, San Antonio, Texas
  - Investigational Site Number 840035, Richmond, Virginia
  - Investigational Site Number 840054, Everett, Washington
  - Investigational Site Number 840033, Tacoma, Washington
- Argentina (11):
  - Investigational Site Number 032004, Buenos Aires
  - Investigational Site Number 032003, Buenos Aires
  - Investigational Site Number 032008, Caba
  - Investigational Site Number 032010, Caba
  - Investigational Site Number 032001, Caba
  - Investigational Site Number 032002, La Plata
  - Investigational Site Number 032005, Rosario
  - Investigational Site Number 032006, Rosario
  - Investigational Site Number 032007, Rosario
  - Investigational Site Number 032009, San Miguel de Tucumán
  - Investigational Site Number 032012, Santa Fe
- Australia (8):
  - Investigational Site Number 036004, Adelaide
  - Investigational Site Number 036002, Brisbane
  - Investigational Site Number 036005, Campbelltown
  - Investigational Site Number 036001, Clayton
  - Investigational Site Number 036008, Frankston
  - Investigational Site Number 036003, Nedlands
  - Investigational Site Number 036009, Prahran
  - Investigational Site Number 036006, Woolloongabba
- Chile (11):
  - Investigational Site Number 152007, Quillota
  - Investigational Site Number 152011, Santiago
  - Investigational Site Number 152001, Santiago
  - Investigational Site Number 152002, Santiago
  - Investigational Site Number 152014, Santiago
  - Investigational Site Number 152003, Santiago
  - Investigational Site Number 152005, Santiago
  - Investigational Site Number 152012, Santiago
  - Investigational Site Number 152013, Santiago
  - Investigational Site Number 152008, Talca
  - Investigational Site Number 152006, Viña del Mar
- France (11):
  - Investigational Site Number 250009, Brest
  - Investigational Site Number 250004, Grenoble
  - Investigational Site Number 250010, Lille
  - Investigational Site Number 250006, Lyon
  - Investigational Site Number 250001, Marseille
  - Investigational Site Number 250002, Montpellier
  - Investigational Site Number 250005, Nantes
  - Investigational Site Number 250007, Nîmes
  - Investigational Site Number 250003, Pessac
  - Investigational Site Number 250008, Strasbourg
  - Investigational Site Number 250011, Vernon
- Italy (10):
  - Investigational Site Number 380010, Ancona
  - Investigational Site Number 380009, Catania
  - Investigational Site Number 380004, Ferrara
  - Investigational Site Number 380002, Florence
  - Investigational Site Number 380008, Foggia
  - Investigational Site Number 380003, Modena
  - Investigational Site Number 380007, Padua
  - Investigational Site Number 380001, Pisa
  - Investigational Site Number 380005, Torino
  - Investigational Site Number 380006, Verona
- Japan (40):
  - Investigational Site Number 392009, Asahi-Shi
  - Investigational Site Number 392037, Chiyoda-Ku
  - Investigational Site Number 392007, Chuoh-Ku
  - Investigational Site Number 392002, Chūōku
  - Investigational Site Number 392012, Edogawa-Ku
  - Investigational Site Number 392017, Fukuoka
  - Investigational Site Number 392021, Fukuyama-Shi
  - Investigational Site Number 392030, Habikino-Shi
  - Investigational Site Number 392004, Himeji-Shi
  - Investigational Site Number 392032, Hirakata-Shi
  - Investigational Site Number 392013, Iizuka-Shi
  - Investigational Site Number 392042, Isesaki-Shi
  - Investigational Site Number 392026, Itabashi-Ku
  - Investigational Site Number 392023, Kanazawa
  - Investigational Site Number 392001, Kitakyushu-Shi
  - Investigational Site Number 392022, Kiyose-Shi
  - Investigational Site Number 392025, Kobe
  - Investigational Site Number 392040, Kodaira-Shi
  - Investigational Site Number 392044, Kokubunji-Shi
  - Investigational Site Number 392010, Kurashiki-Shi
  - Investigational Site Number 392036, Kyoto
  - Investigational Site Number 392041, Nagaoka-Shi
  - Investigational Site Number 392020, Naka-Gun
  - Investigational Site Number 392015, Nakano
  - Investigational Site Number 392005, Naruto-Shi
  - Investigational Site Number 392043, Ohta-Shi
  - Investigational Site Number 392019, Sagamihara-Shi
  - Investigational Site Number 392011, Sakaide-Shi
  - Investigational Site Number 392024, Sakaishi
  - Investigational Site Number 392008, Sapporo
  - Investigational Site Number 392034, Sapporo
  - Investigational Site Number 392038, Setagaya-Ku
  - Investigational Site Number 392028, Sumida-Ku
  - Investigational Site Number 392006, Tomakomai-Shi
  - Investigational Site Number 392003, Toride-Shi
  - Investigational Site Number 392029, Tsu
  - Investigational Site Number 392018, Tsukubo-Gun
  - Investigational Site Number 392045, Uruma
  - Investigational Site Number 392014, Yokohama
  - Investigational Site Number 392035, Yokohama
- Mexico (5):
  - Investigational Site Number 484006, Chihuahua City
  - Investigational Site Number 484005, Distrito Federal
  - Investigational Site Number 484001, Guadalajara
  - Investigational Site Number 484004, Mexico City
  - Investigational Site Number 484003, Monterrey
- New Zealand (2):
  - Investigational Site Number 554001, Dunedin
  - Investigational Site Number 554002, Wellington
- Poland (7):
  - Investigational Site Number 616006, Bialystok
  - Investigational Site Number 616004, Gdansk
  - Investigational Site Number 616003, Gdansk
  - Investigational Site Number 616007, Krakow
  - Investigational Site Number 616001, Lodz
  - Investigational Site Number 616005, Lodz
  - Investigational Site Number 616008, Warsaw
- Russia (10):
  - Investigational Site Number 643003, Moscow
  - Investigational Site Number 643002, Moscow
  - Investigational Site Number 643007, Moscow
  - Investigational Site Number 643012, Moscow
  - Investigational Site Number 643001, Moscow
  - Investigational Site Number 643006, Novosibirsk
  - Investigational Site Number 643010, Saint Petersburg
  - Investigational Site Number 643011, Saint Petersburg
  - Investigational Site Number 643009, Saint Petersburg
  - Investigational Site Number 643008, Yaroslavl
- South Africa (2):
  - Investigational Site Number 710001, Cape Town
  - Investigational Site Number 710002, Cape Town
- South Korea (5):
  - Investigational Site Number 410002, Bucheon-si
  - Investigational Site Number 410003, Cheongju-si
  - Investigational Site Number 410004, Seoul
  - Investigational Site Number 410005, Seoul
  - Investigational Site Number 410001, Suwon
- Spain (7):
  - Investigational Site Number 724005, Barcelona
  - Investigational Site Number 724002, Barcelona
  - Investigational Site Number 724001, Barcelona
  - Investigational Site Number 724004, Cáceres
  - Investigational Site Number 724006, Pozuelo de Alarcón
  - Investigational Site Number 724003, Sabadell
  - Investigational Site Number 724007, Sant Boi de Llobregat
- Turkey (Türkiye) (10):
  - Investigational Site Number 792011, Amasya
  - Investigational Site Number 792002, Ankara
  - Investigational Site Number 792008, Bursa
  - Investigational Site Number 792007, Istanbul
  - Investigational Site Number 792001, Istanbul
  - Investigational Site Number 792004, Istanbul
  - Investigational Site Number 792003, Istanbul
  - Investigational Site Number 792005, Izmir
  - Investigational Site Number 792013, Kırıkkale
  - Investigational Site Number 792006, Mersin
- Ukraine (12):
  - Investigational Site Number 804016, Donetsk
  - Investigational Site Number 804001, Kharkiv
  - Investigational Site Number 804004, Kyiv
  - Investigational Site Number 804003, Kyiv
  - Investigational Site Number 804008, Kyiv
  - Investigational Site Number 804018, Kyiv
  - Investigational Site Number 804020, Kyiv
  - Investigational Site Number 804006, Odesa
  - Investigational Site Number 804002, Poltava
  - Investigational Site Number 804019, Vinnytsia
  - Investigational Site Number 804015, Yalta
  - Investigational Site Number 804012, Zaporizhzhya

REFERENCES:
- [Result] Wenzel S, Castro M, Corren J, Maspero J, Wang L, Zhang B, Pirozzi G, Sutherland ER, Evans RR, Joish VN, Eckert L, Graham NM, Stahl N, Yancopoulos GD, Louis-Tisserand M, Teper A. Dupilumab efficacy and safety in adults with uncontrolled persistent asthma despite use of medium-to-high-dose inhaled corticosteroids plus a long-acting beta2 agonist: a randomised double-blind placebo-controlled pivotal phase 2b dose-ranging trial. Lancet. 2016 Jul 2;388(10039):31-44. doi: 10.1016/S0140-6736(16)30307-5. Epub 2016 Apr 27. PMID 27130691
- [Derived] Pavord ID, Bourdin A, Papi A, Domingo C, Corren J, Altincatal A, Radwan A, Pandit-Abid N, Jacob-Nara JA, Deniz Y, Rowe PJ, Laws E, Lederer DJ, Hardin M. Dupilumab sustains efficacy in patients with moderate-to-severe type 2 asthma regardless of inhaled corticosteroids dose. Allergy. 2023 Nov;78(11):2921-2932. doi: 10.1111/all.15792. Epub 2023 Jul 11. PMID 37431558
- [Derived] Wechsler ME, Klion AD, Paggiaro P, Nair P, Staumont-Salle D, Radwan A, Johnson RR, Kapoor U, Khokhar FA, Daizadeh N, Chen Z, Laws E, Ortiz B, Jacob-Nara JA, Mannent LP, Rowe PJ, Deniz Y. Effect of Dupilumab on Blood Eosinophil Counts in Patients With Asthma, Chronic Rhinosinusitis With Nasal Polyps, Atopic Dermatitis, or Eosinophilic Esophagitis. J Allergy Clin Immunol Pract. 2022 Oct;10(10):2695-2709. doi: 10.1016/j.jaip.2022.05.019. Epub 2022 May 28. PMID 35636689
- [Derived] Bourdin A, Papi AA, Corren J, Virchow JC, Rice MS, Deniz Y, Djandji M, Rowe P, Pavord ID. Dupilumab is effective in type 2-high asthma patients receiving high-dose inhaled corticosteroids at baseline. Allergy. 2021 Jan;76(1):269-280. doi: 10.1111/all.14611. Epub 2020 Oct 21. PMID 33010038
- [Derived] Maspero JF, Katelaris CH, Busse WW, Castro M, Corren J, Chipps BE, Peters AT, Pavord ID, Ford LB, Sher L, Rabe KF, Rice MS, Rowe P, Lu Y, Harel S, Jagerschmidt A, Khan AH, Kamat S, Pirozzi G, Amin N, Ruddy M, Graham NMH, Mannent LP, Teper A. Dupilumab Efficacy in Uncontrolled, Moderate-to-Severe Asthma with Self-Reported Chronic Rhinosinusitis. J Allergy Clin Immunol Pract. 2020 Feb;8(2):527-539.e9. doi: 10.1016/j.jaip.2019.07.016. Epub 2019 Jul 24. PMID 31351189
- [Derived] Corren J, Castro M, Ford LB, Bernstein JA, Jayawardena S, Maroni J, Rowe P, Amin N, Pirozzi G, Graham NMH, Khan A, Eckert L, Teper A. Dupilumab improves asthma outcomes irrespective of frequency of previous asthma exacerbation history. Ann Allergy Asthma Immunol. 2019 Aug;123(2):222-224.e1. doi: 10.1016/j.anai.2019.04.028. Epub 2019 May 8. No abstract available. PMID 31075309
- [Derived] Corren J, Castro M, Chanez P, Fabbri L, Joish VN, Amin N, Graham NMH, Mastey V, Abbe A, Taniou C, Mahajan P, Teper A, Pirozzi G, Eckert L. Dupilumab improves symptoms, quality of life, and productivity in uncontrolled persistent asthma. Ann Allergy Asthma Immunol. 2019 Jan;122(1):41-49.e2. doi: 10.1016/j.anai.2018.08.005. Epub 2018 Aug 21. PMID 30138668
- [Derived] Weinstein SF, Katial R, Jayawardena S, Pirozzi G, Staudinger H, Eckert L, Joish VN, Amin N, Maroni J, Rowe P, Graham NMH, Teper A. Efficacy and safety of dupilumab in perennial allergic rhinitis and comorbid asthma. J Allergy Clin Immunol. 2018 Jul;142(1):171-177.e1. doi: 10.1016/j.jaci.2017.11.051. Epub 2018 Jan 31. PMID 29355679

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 201 sites in 16 countries. A total of 1532 participants were screened between June 2013 and June 2014, of which, 776 participants were randomized at 174 sites in 15 countries. 756 participants were screen failures mainly due to exclusion criteria met and inclusion criteria not met.
Pre-assignment Details: Randomization was stratified using blood eosinophils count (eosinophils >=0.3 Giga/L [G/L]; eosinophils 0.2 to 0.299 G/L; eosinophils<0.2 G/L) and country. Assignment was done by Interactive Voice/Web Response System (1:1:1:1:1) for Placebo and Dupilumab (300 mg every 2 weeks [q2w]; 200 mg q2w; 300 mg every 4 week [q4w] and 200 mg q4w).
Groups:
- Placebo q2w: 2 subcutaneous injections of Placebo (for Dupilumab) as a loading dose on Day 1 (Week 1) followed by a single injection q2w from Week 2 to Week 22 added to stable inhaled corticosteroid/ long-acting beta-agonist (ICS/LABA) therapy. Salbutamol/albuterol or Levosalbutamol/levalbuterol was given as reliever medication.
- Dupilumab 300 mg q2w: 2 subcutaneous injections of Dupilumab 300 mg (for a total of 600 mg) as a loading dose on Day 1 (Week 1), followed by a single 300 mg injection q2w from Week 2 to Week 22 added to stable ICS/LABA therapy. Salbutamol/albuterol or Levosalbutamol/levalbuterol was given as reliever medication.
Period: Overall Study
Arm/Group | Placebo q2w | Dupilumab 300 mg q2w | Dupilumab 200 mg q2w | Dupilumab 300 mg q4w | Dupilumab 200 mg q4w
Started (Started = Randomized) | 158 | 157 | 150 | 157 | 154
Treated | 158 | 156 | 148 | 157 | 150
Completed 12-week Study Treatment | 153 | 149 | 141 | 146 | 143
Completed (Completed = Completed study treatment period.) | 146 | 149 | 137 | 142 | 135
Not Completed | 12 | 8 | 13 | 15 | 19
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 0
Not completed — Poor compliance to protocol | 3 | 0 | 2 | 0 | 0
Not completed — Adverse Event | 5 | 4 | 6 | 10 | 7
Not completed — Randomized but not treated | 0 | 1 | 2 | 0 | 4
Not completed — Other than specified above | 3 | 3 | 3 | 5 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo q2w | Dupilumab 300 mg q2w | Dupilumab 200 mg q2w | Dupilumab 300 mg q4w | Dupilumab 200 mg q4w | Total
Number analyzed (Participants) | 158 | 157 | 150 | 157 | 154 | 776
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (12.7) | 47.5 (12.4) | 51 (13.4) | 47.9 (13.1) | 47.9 (13.1) | 48.6 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 103 | 96 | 100 | 87 | 490
  Male | 54 | 54 | 54 | 57 | 67 | 286
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 0 | 1
  Asian | 25 | 22 | 25 | 23 | 20 | 115
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 0 | 1
  Black or African American | 9 | 5 | 9 | 12 | 7 | 42
  White | 119 | 129 | 114 | 120 | 125 | 607
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 1 | 1 | 1 | 2 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic Or Latino | 31 | 29 | 29 | 33 | 26 | 148
  Not Hispanic Or Latino | 127 | 128 | 121 | 124 | 128 | 628
Number of Participants According to Blood Eosinophil Count [Count of Participants; unit: Participants]
  <0.3 G/L | 90 | 93 | 85 | 91 | 92 | 451
  >=0.3 G/L | 68 | 64 | 65 | 66 | 62 | 325

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1) at Week 12: High Eosinophils -Intent to Treat (HEos-ITT) Population
Description: FEV1 was the volume of air exhaled in the first second of a forced expiration as measured by spirometer.
Time Frame: Baseline, Week 12
Population: HEos-ITT population: subset of intent to treat (ITT) population (defined as randomized population analyzed according to the treatment group allocated by randomization, regardless of whether the treatment was actually received) which included participants with baseline blood eosinophils >=0.3 G/L.
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | Placebo q2w | Dupilumab 300 mg q2w | Dupilumab 200 mg q2w | Dupilumab 300 mg q4w | Dupilumab 200 mg q4w
Number analyzed (Participants) | 68 | 64 | 65 | 66 | 62
liter
  Baseline | 1.86 (0.68) | 1.77 (0.5) | 1.8 (0.52) | 1.87 (0.6) | 1.8 (0.49)
  Week 12: number analyzed (Participants) | 58 | 59 | 57 | 55 | 53
  Week 12 | 2.13 (0.78) | 2.12 (0.54) | 2.26 (0.68) | 2.26 (0.70) | 2.09 (0.54)
  Change from baseline at Week 12: number analyzed (Participants) | 58 | 59 | 57 | 55 | 53
  Change from baseline at Week 12 | 0.18 (0.38) | 0.36 (0.46) | 0.45 (0.40) | 0.35 (0.43) | 0.26 (0.47)
Statistical Analysis 1: Comparison: Placebo q2w vs Dupilumab 300 mg q2w; Analysis was performed using mixed effect model with repeated measures (MMRM) approach including available FEV1 data from baseline to Week 12 and treatment group as a factor. A step-down procedure was used to strongly control the overall type I error rate for testing multiple doses against placebo. The hierarchy was 300 mg q2w, 200 mg q2w, 300 mg q4w, and 200 mg q4w; Test type: Superiority; p = 0.0063, Mixed Models Analysis — Threshold for significance at 0.05; Least Square (LS) Mean Difference = 0.21, 95% CI 2-sided [0.06 to 0.36] — Dupilumab 300 mg q2w vs. Placebo q2w
Statistical Analysis 2: Comparison: Placebo q2w vs Dupilumab 200 mg q2w; Test type: Superiority; p = 0.0008, Mixed Models Analysis — Threshold for significance at 0.05; LS Mean Difference = 0.26, 95% CI 2-sided [0.11 to 0.40] — Dupilumab 200 mg q2w vs. Placebo q2w
Statistical Analysis 3: Comparison: Placebo q2w vs Dupilumab 300 mg q4w; Test type: Superiority; p = 0.0212, Mixed Models Analysis — Threshold for significance at 0.05; LS Mean Difference = 0.17, 95% CI 2-sided [0.03 to 0.32] — Dupilumab 300 mg q4w vs. Placebo q2w
Statistical Analysis 4: Comparison: Placebo q2w vs Dupilumab 200 mg q4w; Test type: Superiority; p = 0.2774, Mixed Models Analysis — Threshold for significance at 0.05; LS Mean Difference = 0.08, 95% CI 2-sided [-0.07 to 0.23] — Dupilumab 200 mg q4w vs. Placebo q2w

2. Primary Outcome: Absolute Change From Baseline in FEV1 at Week 12: ITT Population
Description: FEV1 was the volume of air exhaled in the first second of a forced expiration as measured by spirometer.
Time Frame: Baseline, Week 12
Population: ITT population.
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | Placebo q2w | Dupilumab 300 mg q2w | Dupilumab 200 mg q2w | Dupilumab 300 mg q4w | Dupilumab 200 mg q4w
Number analyzed (Participants) | 158 | 157 | 150 | 157 | 154
liter
  Baseline | 1.82 (0.55) | 1.85 (0.53) | 1.79 (0.52) | 1.86 (0.57) | 1.88 (0.54)
  Week 12: number analyzed (Participants) | 129 | 146 | 136 | 134 | 134
  Week 12 | 2.01 (0.69) | 2.12 (0.59) | 2.12 (0.68) | 2.14 (0.69) | 2.07 (0.63)
  Change from baseline at Week 12: number analyzed (Participants) | 129 | 146 | 136 | 134 | 134
  Change from baseline at Week 12 | 0.13 (0.37) | 0.26 (0.39) | 0.32 (0.38) | 0.24 (0.4) | 0.20 (0.41)
Statistical Analysis 1: Comparison: Placebo q2w vs Dupilumab 300 mg q2w; Analysis was performed using MMRM approach including available FEV1 data from baseline to Week 12 and treatment group as a factor. A step-down procedure was used to strongly control the overall type I error rate for testing multiple doses against placebo. The hierarchy was 300 mg q2w, 200 mg q2w, 300 mg q4w and 200 mg q4w; Test type: Superiority; p = 0.0002, Mixed Models Analysis — Threshold for significance at 0.05; LS Mean Difference = 0.16, 95% CI 2-sided [0.08 to 0.25] — Dupilumab 300 mg q2w vs. Placebo q2w
Statistical Analysis 2: Comparison: Placebo q2w vs Dupilumab 200 mg q2w; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05; LS Mean Difference = 0.2, 95% CI 2-sided [0.011 to 0.28] — Dupilumab 200 mg q2w vs. Placebo q2w
Statistical Analysis 3: Comparison: Placebo q2w vs Dupilumab 300 mg q4w; Test type: Superiority; p = 0.0048, Mixed Models Analysis — Threshold for significance at 0.05; LS Mean Difference = 0.12, 95% CI 2-sided [0.04 to 0.21] — Dupilumab 300 mg q4w vs. Placebo q2w
Statistical Analysis 4: Comparison: Placebo q2w vs Dupilumab 200 mg q4w; Test type: Superiority; p = 0.0304, Mixed Models Analysis — Threshold for significance at 0.05; LS Mean Difference = 0.10, 95% CI 2-sided [0.01 to 0.18] — Dupilumab 200 mg q4w vs. Placebo q2w

3. Secondary Outcome: Percent Change From Baseline in FEV1 at Week 12: HEos-ITT Population
Description: FEV1 was the volume of air exhaled in the first second of a forced expiration as measured by spirometer.
Time Frame: Baseline, Week 12
Population: HEos-ITT population. Here 'overall number of participants analyzed' signifies participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo q2w | Dupilumab 300 mg q2w | Dupilumab 200 mg q2w | Dupilumab 300 mg q4w | Dupilumab 200 mg q4w
Number analyzed (Participants) | 58 | 59 | 57 | 55 | 53
percent change | 10.07 (19.65) | 25.29 (36.15) | 27.42 (25.68) | 20.68 (24.86) | 18.07 (29.18)

4. Secondary Outcome: Percent Change From Baseline in FEV1 at Week 12: ITT Population
Description: FEV1 was the volume of air exhaled in the first second of a forced expiration as measured by spirometer.
Time Frame: Baseline, Week 12
Population: ITT population. Here 'overall number of participants analyzed' signifies participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo q2w | Dupilumab 300 mg q2w | Dupilumab 200 mg q2w | Dupilumab 300 mg q4w | Dupilumab 200 mg q4w
Number analyzed (Participants) | 129 | 146 | 136 | 134 | 134
percent change | 7.04 (19.26) | 16.64 (27.78) | 19.15 (23.53) | 13.55 (23.01) | 13.04 (24.21)

5. Secondary Outcome: Annualized Event Rate of Severe Exacerbation During The Treatment Period: HEos-ITT Population
Description: A severe exacerbation was defined as a deterioration of asthma requiring: use of systemic corticosteroids for >=3 days; or hospitalization or emergency room visit because of asthma, requiring systemic corticosteroids. Annualized event rate was the total number of exacerbations that occurred during the treatment period divided by the total number of participant-years treated.
Time Frame: Baseline to Week 24
Population: HEos-ITT population. Here 'overall number of participants analyzed' signifies participants of the HEos-ITT population who were treated.
Measure: Number (95% Confidence Interval); unit: exacerbation per participant-year
Arm/Group | Placebo q2w | Dupilumab 300 mg q2w | Dupilumab 200 mg q2w | Dupilumab 300 mg q4w | Dupilumab 200 mg q4w
Number analyzed (Participants) | 68 | 64 | 64 | 66 | 59
exacerbation per participant-year | 1.044 [0.572 to 1.904] | 0.201 [0.078 to 0.517] | 0.30 [0.133 to 0.678] | 0.678 [0.356 to 1.29] | 0.358 [0.158 to 0.809]

6. Secondary Outcome: Annualized Event Rate of Severe Exacerbation During The Treatment Period: ITT Population
Description: as for outcome 5
Time Frame: Baseline to Week 24
Population: ITT population. Here 'overall number of participants analyzed' signifies participants of the ITT population who were treated.
Measure: Number (95% Confidence Interval); unit: exacerbation per participant-year
Arm/Group | Placebo q2w | Dupilumab 300 mg q2w | Dupilumab 200 mg q2w | Dupilumab 300 mg q4w | Dupilumab 200 mg q4w
Number analyzed (Participants) | 158 | 156 | 148 | 157 | 150
exacerbation per participant-year | 0.897 [0.619 to 1.30] | 0.265 [0.157 to 0.445] | 0.269 [0.157 to 0.461] | 0.599 [0.369 to 0.907] | 0.415 [0.26 to 0.664]

7. Secondary Outcome: Time to First Severe Exacerbation: Kaplan-Meier Estimates at Week 12 and 24: HEos-ITT Population
Description: The time to first severe exacerbation was defined as the time from the date of first dose to the date of the first severe exacerbation event. For participants who had no severe exacerbation on or before last dose date + 14 days, it was censored at the date of last dose date + 14 days. The median time to first severe exacerbation was not estimated because the number of severe exacerbations was too low in the Dupilumab arms. Therefore, alternative Kaplan-Meier statistics, the probability of severe exacerbation at Week 12 and 24, are presented as the descriptive measure statistics.
Time Frame: Baseline up to Week 24
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: probability of Severe Exacerbation
Arm/Group | Placebo q2w | Dupilumab 300 mg q2w | Dupilumab 200 mg q2w | Dupilumab 300 mg q4w | Dupilumab 200 mg q4w
Number analyzed (Participants) | 68 | 64 | 64 | 66 | 59
probability of Severe Exacerbation
  Probability at Week 12 | 0.21 [0.122 to 0.314] | 0.082 [0.03 to 0.167] | 0.082 [0.03 to 0.167] | 0.094 [0.038 to 0.181] | 0.052 [0.014 to 0.13]
  Probability at Week 24 | 0.287 [0.184 to 0.398] | 0.116 [0.051 to 0.21] | 0.082 [0.03 to 0.167] | 0.175 [0.093 to 0.278] | 0.125 [0.055 to 0.226]

8. Secondary Outcome: Time to First Severe Exacerbation: Kaplan-Meier Estimates at Week 12 and 24: ITT Population
Description: as for outcome 7
Time Frame: Baseline up to Week 24
Population: ITT population. Here 'overall number of participants analyzed' signifies participants of ITT population who were treated.
Measure: Number (95% Confidence Interval); unit: probability of Severe Exacerbation
Arm/Group | Placebo q2w | Dupilumab 300 mg q2w | Dupilumab 200 mg q2w | Dupilumab 300 mg q4w | Dupilumab 200 mg q4w
Number analyzed (Participants) | 158 | 156 | 148 | 157 | 150
probability of Severe Exacerbation
  Probability at Week 12 | 0.207 [0.147 to 0.274] | 0.092 [0.053 to 0.145] | 0.07 [0.036 to 0.119] | 0.112 [0.068 to 0.168] | 0.075 [0.04 to 0.125]
  Probability at Week 24 | 0.266 [0.199 to 0.338] | 0.112 [0.068 to 0.169] | 0.091 [0.051 to 0.145] | 0.195 [0.136 to 0.262] | 0.16 [0.106 to 0.225]

9. Secondary Outcome: Annualized Event Rate of Loss of Asthma Control (LOAC) During The Treatment Period: HEos-ITT Population
Description: LOAC was defined as any of the following: >=6 additional reliever puffs of salbutamol/albuterol or levosalbutamol/levalbuterol in a 24-hour period (compared to baseline) on 2 consecutive days; increase in inhaled corticosteroid (ICS) >=4 times the dose at randomization; use of systemic corticosteroids for >=3 days; hospitalization or emergency room visit because of asthma, requiring systemic corticosteroids. Annualized event rate was the total number of LOAC that occurred during the treatment period divided by the total number of participant-years treated.
Time Frame: Baseline to Week 24
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: LOAC per participant-year
Arm/Group | Placebo q2w | Dupilumab 300 mg q2w | Dupilumab 200 mg q2w | Dupilumab 300 mg q4w | Dupilumab 200 mg q4w
Number analyzed (Participants) | 68 | 64 | 64 | 66 | 59
LOAC per participant-year | 1.312 [0.804 to 2.142] | 0.322 [0.153 to 0.677] | 0.446 [0.231 to 0.864] | 0.788 [0.458 to 1.355] | 0.424 [0.212 to 0.851]

10. Secondary Outcome: Annualized Event Rate of LOAC During The Treatment Period: ITT Population
Description: LOAC was defined as any of the following: >=6 additional reliever puffs of salbutamol/albuterol or levosalbutamol/levalbuterol in a 24-hour period (compared to baseline) on 2 consecutive days; increase in ICS >=4 times the dose at randomization; use of systemic corticosteroids for >=3 days; hospitalization or emergency room visit because of asthma, requiring systemic corticosteroids. Annualized event rate was the total number of LOAC that occurred during the treatment period divided by the total number of participant-years treated.
Time Frame: Baseline to Week 24
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: LOAC per participant-year
Arm/Group | Placebo q2w | Dupilumab 300 mg q2w | Dupilumab 200 mg q2w | Dupilumab 300 mg q4w | Dupilumab 200 mg q4w
Number analyzed (Participants) | 158 | 156 | 148 | 157 | 150
LOAC per participant-year | 1.107 [0.801 to 1.53] | 0.326 [0.206 to 0.515] | 0.347 [0.217 to 0.555] | 0.73 [0.508 to 1.048] | 0.563 [0.378 to 0.839]

11. Secondary Outcome: Time to First LOAC Event: Kaplan-Meier Estimates at Week 12 and Week 24: HEos-ITT Population
Description: The time to first LOAC event was defined as the time from the date of first dose to the date of the first LOAC event. For participants who had no LOAC event on or before last dose date + 14 days, it was censored at the date of last dose date + 14 days. The median time to first LOAC was not estimated because the number of LOAC was too low in the Dupilumab arms. Therefore, alternative Kaplan-Meier statistics, the probability of LOAC at Week 12 and 24, are presented as the descriptive measure statistics.
Time Frame: Baseline up to Week 24
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: probability of LOAC
Arm/Group | Placebo q2w | Dupilumab 300 mg q2w | Dupilumab 200 mg q2w | Dupilumab 300 mg q4w | Dupilumab 200 mg q4w
Number analyzed (Participants) | 68 | 64 | 64 | 66 | 59
probability of LOAC
  Probability at Week 12 | 0.30 [0.195 to 0.411] | 0.115 [0.05 to 0.208] | 0.113 [0.05 to 0.206] | 0.126 [0.059 to 0.22] | 0.052 [0.014 to 0.13]
  Probability at Week 24 | 0.392 [0.275 to 0.507] | 0.166 [0.085 to 0.269] | 0.113 [0.05 to 0.206] | 0.207 [0.117 to 0.314] | 0.162 [0.079 to 0.269]

12. Secondary Outcome: Time to First LOAC Event: Kaplan-Meier Estimates at Week 12 and Week 24: ITT Population
Description: as for outcome 11
Time Frame: Baseline up to Week 24
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: probability of LOAC
Arm/Group | Placebo q2w | Dupilumab 300 mg q2w | Dupilumab 200 mg q2w | Dupilumab 300 mg q4w | Dupilumab 200 mg q4w
Number analyzed (Participants) | 158 | 156 | 148 | 157 | 150
probability of LOAC
  Probability at Week 12 | 0.258 [0.192 to 0.329] | 0.112 [0.068 to 0.168] | 0.09 [0.051 to 0.144] | 0.145 [0.095 to 0.206] | 0.096 [0.055 to 0.15]
  Probability at Week 24 | 0.338 [0.265 to 0.413] | 0.146 [0.095 to 0.207] | 0.112 [0.067 to 0.169] | 0.242 [0.177 to 0.314] | 0.209 [0.147 to 0.279]

13. Secondary Outcome: Change From Baseline in Morning Asthma Symptom Score at Week 12: HEos-ITT Population
Description: Morning asthma symptom score was determined using AM (ante meridiem) symptom scoring system which evaluated participant's overall asthma symptoms experienced during the night. It ranged from 0 to 4 as: 0 = No asthma symptoms, slept through the night, 1= Slept well, but some complaints in the morning, no night-time awakenings, 2= Woke up once because of asthma (including early awakening), 3= Woke up several times because of asthma (including early awakening), 4= Bad night, awake most of the night because of asthma.
Time Frame: Baseline, Week 12
Population: HEos-ITT population.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo q2w | Dupilumab 300 mg q2w | Dupilumab 200 mg q2w | Dupilumab 300 mg q4w | Dupilumab 200 mg q4w
Number analyzed (Participants) | 68 | 64 | 65 | 66 | 62
scores on a scale
  Baseline | 1.15 (0.82) | 1.45 (0.81) | 1.22 (0.81) | 1.31 (0.72) | 1.18 (0.82)
  Week 12: number analyzed (Participants) | 62 | 59 | 58 | 61 | 56
  Week 12 | 0.83 (0.66) | 0.78 (0.88) | 0.70 (0.69) | 0.70 (0.78) | 0.63 (0.62)
  Change from baseline at Week 12: number analyzed (Participants) | 62 | 59 | 58 | 61 | 56
  Change from baseline at Week 12 | -0.29 (0.70) | -0.66 (0.67) | -0.55 (0.75) | -0.57 (0.63) | -0.57 (0.60)

14. Secondary Outcome: Change From Baseline in Morning Asthma Symptom Score at Week 12: ITT Population
Description: Morning asthma symptom score was determined using AM symptom scoring system which evaluated participant's overall asthma symptoms experienced during the night. It ranged from 0 to 4 as: 0 = No asthma symptoms, slept through the night, 1= Slept well, but some complaints in the morning, no night-time awakenings, 2= Woke up once because of asthma (including early awakening), 3= Woke up several times because of asthma (including early awakening), 4= Bad night, awake most of the night because of asthma.
Time Frame: Baseline, Week 12
Population: ITT population.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo q2w | Dupilumab 300 mg q2w | Dupilumab 200 mg q2w | Dupilumab 300 mg q4w | Dupilumab 200 mg q4w
Number analyzed (Participants) | 158 | 157 | 150 | 157 | 154
scores on a scale
  Baseline | 1.17 (0.79) | 1.25 (0.78) | 1.24 (0.81) | 1.33 (0.78) | 1.29 (0.82)
  Week 12: number analyzed (Participants) | 143 | 148 | 138 | 148 | 140
  Week 12 | 0.90 (0.67) | 0.82 (0.79) | 0.79 (0.77) | 0.80 (0.73) | 0.72 (0.68)
  Change from baseline at Week 12: number analyzed (Participants) | 143 | 148 | 138 | 148 | 140
  Change from baseline at Week 12 | -0.23 (0.70) | -0.43 (0.70) | -0.46 (0.75) | -0.52 (0.65) | -0.54 (0.64)

15. Secondary Outcome: Change From Baseline in Evening Asthma Symptom Score at Week 12: HEos-ITT Population
Description: Evening asthma symptom score was determined using PM (post meridiem) symptom scoring system which evaluated participant's overall asthma symptoms experienced during the day. It ranged from 0 to 4 as: 0=very well, no asthma symptoms, 1=one episode of wheezing, cough, or breathlessness, 2=more than one episode of wheezing, cough, or breathlessness without interference of normal activities, 3=wheezing, cough, or breathlessness most of the day, which interfered to some extent with normal activities, 4=asthma very bad, unable to carry out daily activities as usual.
Time Frame: Baseline, Week 12
Population: HEos ITT population.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo q2w | Dupilumab 300 mg q2w | Dupilumab 200 mg q2w | Dupilumab 300 mg q4w | Dupilumab 200 mg q4w
Number analyzed (Participants) | 68 | 64 | 65 | 66 | 62
scores on a scale
  Baseline | 1.33 (0.83) | 1.72 (0.89) | 1.46 (0.73) | 1.52 (0.72) | 1.39 (0.87)
  Week 12: number analyzed (Participants) | 62 | 59 | 58 | 61 | 56
  Week 12 | 0.95 (0.71) | 0.88 (0.91) | 0.89 (0.79) | 0.76 (0.84) | 0.69 (0.68)
  Change from baseline at Week 12: number analyzed (Participants) | 62 | 59 | 58 | 61 | 56
  Change from baseline at Week 12 | -0.35 (0.71) | -0.84 (0.87) | -0.62 (0.70) | -0.73 (0.77) | -0.69 (0.70)

16. Secondary Outcome: Change From Baseline in Evening Asthma Symptom Score at Week 12: ITT Population
Description: Evening asthma symptom score was determined using PM symptom scoring system which evaluated participant's overall asthma symptoms experienced during the day. It ranged from 0 to 4 as: 0=very well, no asthma symptoms, 1=one episode of wheezing, cough, or breathlessness, 2=more than one episode of wheezing, cough, or breathlessness without interference of normal activities, 3=wheezing, cough, or breathlessness most of the day, which interfered to some extent with normal activities, 4=asthma very bad, unable to carry out daily activities as usual.
Time Frame: Baseline, Week 12
Population: ITT population.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo q2w | Dupilumab 300 mg q2w | Dupilumab 200 mg q2w | Dupilumab 300 mg q4w | Dupilumab 200 mg q4w
Number analyzed (Participants) | 158 | 157 | 150 | 157 | 154
scores on a scale
  Baseline | 1.32 (0.81) | 1.47 (0.85) | 1.42 (0.79) | 1.50 (0.74) | 1.47 (0.84)
  Week 12: number analyzed (Participants) | 143 | 148 | 136 | 148 | 140
  Week 12 | 1.02 (0.73) | 0.95 (0.88) | 0.95 (0.81) | 0.89 (0.79) | 0.89 (0.81)
  Change from baseline at Week 12: number analyzed (Participants) | 143 | 148 | 136 | 148 | 140
  Change from baseline at Week 12 | -0.27 (0.76) | -0.52 (0.79) | -0.52 (0.80) | -0.59 (0.79) | -0.54 (0.71)

17. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire 5-item Version (ACQ-5) Score at Week 12: HEos-ITT Population
Description: The ACQ-5 has 5 questions, reflecting the top-scoring five asthma symptoms: woken at night by symptoms, wake in the mornings with symptoms, limitation of daily activities, shortness of breath and wheeze. Participants were asked to recall how their asthma had been during the previous week and to respond to each of the five symptom questions on a 7-point scale ranged from 0 (no impairment) to 6 (maximum impairment). ACQ-5 total score was mean of the scores of all 5 questions and, therefore, ranged from 0 (totally controlled) to 6 (severely uncontrolled). Higher score indicated lower asthma control.
Time Frame: Baseline, Week 12
Population: HEos-ITT population.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo q2w | Dupilumab 300 mg q2w | Dupilumab 200 mg q2w | Dupilumab 300 mg q4w | Dupilumab 200 mg q4w
Number analyzed (Participants) | 68 | 64 | 65 | 66 | 62
scores on a scale
  Baseline: number analyzed (Participants) | 68 | 64 | 65 | 66 | 61
  Baseline | 2.55 (0.84) | 2.98 (0.90) | 2.65 (0.74) | 2.69 (0.81) | 2.76 (0.91)
  Week 12: number analyzed (Participants) | 58 | 59 | 56 | 55 | 53
  Week 12 | 1.52 (1.09) | 1.20 (0.96) | 1.20 (0.88) | 1.27 (0.91) | 1.39 (0.94)
  Change from baseline at Week 12: number analyzed (Participants) | 58 | 59 | 56 | 55 | 53
  Change from baseline at Week 12 | -1.03 (0.93) | -1.72 (1.14) | -1.40 (1.03) | -1.39 (1.02) | -1.38 (0.90)

18. Secondary Outcome: Change From Baseline in ACQ-5 Score at Week 12: ITT Population
Description: as for outcome 17
Time Frame: Baseline, Week 12
Population: ITT population.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo q2w | Dupilumab 300 mg q2w | Dupilumab 200 mg q2w | Dupilumab 300 mg q4w | Dupilumab 200 mg q4w
Number analyzed (Participants) | 158 | 157 | 150 | 157 | 154
scores on a scale
  Baseline: number analyzed (Participants) | 158 | 157 | 150 | 157 | 153
  Baseline | 2.69 (0.80) | 2.80 (0.83) | 2.73 (0.82) | 2.70 (0.79) | 2.78 (0.84)
  Week 12: number analyzed (Participants) | 129 | 145 | 134 | 134 | 135
  Week 12 | 1.55 (1.00) | 1.41 (1.02) | 1.38 (0.96) | 1.38 (0.86) | 1.49 (0.98)
  Change from baseline at Week 12: number analyzed (Participants) | 129 | 145 | 134 | 134 | 135
  Change from baseline at Week 12 | -1.11 (0.93) | -1.38 (1.10) | -1.35 (1.05) | -1.32 (1.02) | -1.24 (0.95)

19. Secondary Outcome: Change From Baseline in Asthma Quality of Life Questionnaire (AQLQ) Global Score at Week 12: HEos-ITT Population
Description: The AQLQ is a disease-specific, self-administered quality of life questionnaire designed to measure functional impairments that are most important to participants with asthma. The AQLQ comprises of 32 items in 4 domains: symptoms (12 items), activity limitation (11 items), emotional function (5 items), environmental stimuli (4 items). Each item is scored on a 7-point Likert scale (1=maximal impairment, 7=no impairment). The 32 items of the questionnaire are averaged to produce one overall quality of life score ranging from 1 (severely impaired) to 7 (not impaired at all). Higher scores indicate better quality of life.
Time Frame: Baseline, Week 12
Population: HEos-ITT population.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo q2w | Dupilumab 300 mg q2w | Dupilumab 200 mg q2w | Dupilumab 300 mg q4w | Dupilumab 200 mg q4w
Number analyzed (Participants) | 68 | 64 | 65 | 66 | 62
scores on a scale
  Baseline: number analyzed (Participants) | 68 | 63 | 64 | 66 | 60
  Baseline | 4.16 (1.27) | 3.82 (1.13) | 4.02 (1.15) | 3.99 (1.06) | 3.89 (1.88)
  Week 12: number analyzed (Participants) | 60 | 60 | 58 | 58 | 53
  Week 12 | 5.05 (1.22) | 5.35 (1.21) | 5.41 (1.06) | 5.06 (1.19) | 5.05 (1.29)
  Change from baseline at Week 12: number analyzed (Participants) | 60 | 59 | 57 | 58 | 52
  Change from baseline at Week 12 | 0.80 (1.02) | 1.54 (1.18) | 1.42 (0.97) | 1.08 (0.97) | 1.16 (1.01)

20. Secondary Outcome: Change From Baseline in AQLQ Global Score at Week 12: ITT Population
Description: as for outcome 19
Time Frame: Baseline, Week 12
Population: ITT population.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo q2w | Dupilumab 300 mg q2w | Dupilumab 200 mg q2w | Dupilumab 300 mg q4w | Dupilumab 200 mg q4w
Number analyzed (Participants) | 158 | 157 | 150 | 157 | 154
scores on a scale
  Baseline: number analyzed (Participants) | 156 | 153 | 148 | 157 | 152
  Baseline | 4.12 (1.10) | 3.91 (1.13) | 4.03 (1.15) | 4.02 (1.01) | 4.00 (1.09)
  Week 12: number analyzed (Participants) | 135 | 145 | 136 | 139 | 136
  Week 12 | 5.00 (1.10) | 5.13 (1.22) | 5.22 (1.11) | 5.04 (1.13) | 5.03 (1.12)
  Change from baseline at Week 12: number analyzed (Participants) | 133 | 142 | 134 | 139 | 135
  Change from baseline at Week 12 | 0.86 (0.99) | 1.25 (1.10) | 1.19 (1.05) | 1.03 (1.02) | 0.98 (1.02)

21. Secondary Outcome: Change From Baseline in Number of Inhalations Per Day of Salbutamol/Albuterol or Levosalbutamol/Levalbuterol at Week 12: HEos-ITT Population
Description: Participants might administered salbutamol/albuterol or levosalbutamol/levalbuterol as reliever medication as needed during the study. The number of salbutamol/albuterol or levosalbutamol/levalbuterol inhalations were recorded by the participants in their electronic diary.
Time Frame: Baseline, Week 12
Population: HEos-ITT Population.
Measure: Mean (Standard Deviation); unit: inhalations per day
Arm/Group | Placebo q2w | Dupilumab 300 mg q2w | Dupilumab 200 mg q2w | Dupilumab 300 mg q4w | Dupilumab 200 mg q4w
Number analyzed (Participants) | 68 | 64 | 65 | 66 | 62
inhalations per day
  Baseline | 2.53 (2.77) | 3.61 (3.56) | 3.02 (2.85) | 3.15 (2.70) | 2.42 (2.75)
  Week 12: number analyzed (Participants) | 62 | 59 | 58 | 61 | 56
  Week 12 | 1.88 (2.53) | 2.14 (3.22) | 2.15 (2.67) | 1.85 (2.75) | 1.36 (1.76)
  Change from baseline at Week 12: number analyzed (Participants) | 62 | 59 | 58 | 61 | 56
  Change from baseline at Week 12 | -0.51 (1.74) | -1.47 (2.31) | -0.93 (2.31) | -1.49 (2.37) | -1.01 (2.00)

22. Secondary Outcome: Change From Baseline in Number of Inhalations Per Day of Salbutamol/Albuterol or Levosalbutamol/Levalbuterol at Week 12: ITT Population
Description: as for outcome 21
Time Frame: Baseline, Week 12
Population: ITT population.
Measure: Mean (Standard Deviation); unit: inhalations per day
Arm/Group | Placebo q2w | Dupilumab 300 mg q2w | Dupilumab 200 mg q2w | Dupilumab 300 mg q4w | Dupilumab 200 mg q4w
Number analyzed (Participants) | 158 | 157 | 150 | 157 | 154
inhalations per day
  Baseline | 2.72 (2.73) | 3.25 (3.15) | 2.98 (2.74) | 3.36 (3.43) | 3.01 (2.87)
  Week 12: number analyzed (Participants) | 142 | 148 | 136 | 148 | 140
  Week 12 | 2.20 (2.57) | 2.30 (3.02) | 2.03 (2.46) | 2.09 (2.73) | 1.99 (2.42)
  Change from baseline at Week 12: number analyzed (Participants) | 142 | 148 | 136 | 148 | 140
  Change from baseline at Week 12 | -0.44 (1.75) | -0.95 (2.05) | -0.99 (2.27) | -1.35 (2.84) | -0.92 (2.16)

23. Post Hoc Outcome: Change From Baseline in FEV1 at Week 12: Subset of ITT Population With Baseline Blood Eosinophil <0.3 G/L
Description: FEV1 was the volume of air exhaled in the first second of a forced expiration as measured by spirometer.
Time Frame: Baseline, Week 12
Population: Analysis was performed on subset of ITT population which included participants with baseline blood eosinophil count <0.3 G/L.
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | Placebo q2w | Dupilumab 300 mg q2w | Dupilumab 200 mg q2w | Dupilumab 300 mg q4w | Dupilumab 200 mg q4w
Number analyzed (Participants) | 90 | 93 | 85 | 91 | 92
liter
  Baseline | 1.79 (0.42) | 1.9 (0.55) | 1.79 (0.53) | 1.85 (0.56) | 1.94 (0.56)
  Week 12: number analyzed (Participants) | 71 | 87 | 79 | 79 | 81
  Week 12 | 1.92 (0.61) | 2.12 (0.63) | 2.02 (0.67) | 2.05 (0.68) | 2.06 (0.68)
  Change from baseline at Week 12: number analyzed (Participants) | 71 | 87 | 79 | 79 | 81
  Change from baseline at Week 12 | 0.09 (0.36) | 0.19 (0.31) | 0.23 (0.33) | 0.16 (0.36) | 0.17 (0.36)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected from signature of the informed consent form up to the final visit (Week 40) regardless of seriousness or relationship to investigational product.
Description: Reported AEs and deaths are treatment emergent AEs that developed/worsened and deaths that occurred during 'treatment-emergent period' (from first dose of investigational product injection up to end of 16-week post-treatment period).
Groups:
- Placebo: Participants exposed to Placebo (for Dupilumab) added to stable ICS/LABA therapy (mean exposure of 23 weeks).
- Dupilumab 300 mg q2w: Participants exposed to Dupilumab 300 mg q2w added to stable ICS/LABA therapy (mean exposure of 23 weeks).
- Dupilumab 200 mg q2w: Participants exposed to Dupilumab 200 mg q2w added to stable ICS/LABA therapy (mean exposure of 23 weeks).
- Dupilumab 300 mg q4w: Participants exposed to Dupilumab 300 mg alternating with placebo q2w added to stable ICS/LABA therapy (mean exposure of 23 weeks).
- Dupilumab 200 mg q4w: Participants exposed to Dupilumab 200 mg alternating with placebo q2w added to stable ICS/LABA therapy (mean exposure of 23 weeks).
Arm/Group | Placebo | Dupilumab 300 mg q2w | Dupilumab 200 mg q2w | Dupilumab 300 mg q4w | Dupilumab 200 mg q4w
All-Cause Mortality (participants affected / at risk) | 0/158 | 0/156 | 0/148 | 2/157 | 0/150
Serious Adverse Events (participants affected / at risk) | 9/158 | 13/156 | 10/148 | 16/157 | 6/150
Other Adverse Events (participants affected / at risk) | 88/158 | 95/156 | 81/148 | 96/157 | 74/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=158) | Dupilumab 300 mg q2w (N=156) | Dupilumab 200 mg q2w (N=148) | Dupilumab 300 mg q4w (N=157) | Dupilumab 200 mg q4w (N=150)
Appendicitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Epiglottitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Hypergammaglobulinaemia benign monoclonal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cor pulmonale acute (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 5 | 2 | 2
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Subileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Hepatitis cholestatic (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 2 | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0
Uterine prolapse (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 1 | 0 | 0 | 0
Bone fissure (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Comminuted fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Procedural intestinal perforation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=158) | Dupilumab 300 mg q2w (N=156) | Dupilumab 200 mg q2w (N=148) | Dupilumab 300 mg q4w (N=157) | Dupilumab 200 mg q4w (N=150)
Bronchitis (Infections and infestations) | 16 | 19 | 11 | 11 | 10
Influenza (Infections and infestations) | 5 | 9 | 6 | 13 | 10
Nasopharyngitis (Infections and infestations) | 15 | 16 | 15 | 19 | 9
Pharyngitis (Infections and infestations) | 8 | 5 | 3 | 7 | 3
Sinusitis (Infections and infestations) | 11 | 6 | 5 | 13 | 12
Upper respiratory tract infection (Infections and infestations) | 28 | 20 | 22 | 19 | 22
Headache (Nervous system disorders) | 20 | 17 | 17 | 19 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 11 | 4 | 7 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 6 | 1 | 9 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 3 | 3 | 7 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 12 | 8 | 4 | 7
Injection site erythema (General disorders) | 12 | 34 | 21 | 12 | 13
Injection site oedema (General disorders) | 1 | 8 | 4 | 0 | 2
Injection site pain (General disorders) | 7 | 14 | 7 | 6 | 5
Injection site pruritus (General disorders) | 5 | 12 | 10 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.